CLINICAL TRIAL: NCT00892229
Title: Buccal Versus Vaginal Misoprostol for Cervical Ripening Prior to Surgical Termination of the First Trimester Missed Abortion in Erbil
Brief Title: Buccal Versus Vaginal Misoprostol in Surgical Termination of the First Trimester Missed Abortion in Erbil
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hawler Medical University (Other)
Collaborators: NEGATIVE (Ambiguous)
Responsible Party: Dr. NADA S AMEEN - THE CHAIRWOMEN, IRAQI MEDICAL SPECIALIZATION
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMS - 1769
Record Dates: First submitted 2009-05-01; First posted 2009-05-04 (Estimated); Last update posted 2009-05-04 (Estimated); Status verified 2009-05

CONDITIONS: Missed Abortion
Keywords: First trimester missed abortion; Misoprostol; buccal; vaginal; cervical ripening; first trimester; missed abortion
MeSH Terms: conditions — Abortion, Missed | interventions — Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Buccal Misoprostol (Active Comparator): Group one: 50 patients with first trimester missed abortion received buccal misoprostol
  Interventions: Drug: Misoprostol (given buccally)
- Vaginal Misoprostol (Active Comparator): Group two: 5 patients received vaginal misoprostol
  Interventions: Drug: Misoprostol (given vaginally)
- Buccal and Vaginal Misoprostol (Active Comparator): 50 primiparous and 50 multiparous women: one hundred patients have been administered the medication buccally (25 primigravida and 25 multigravida), and vaginally (25 primigravida and 25 multigravida), three hours before dilation and curettage. They were admitted to the hospital one day before the surgical evacuation, and preparation of cross matched blood done for all recruited subjects.
  Each group was randomly allocated (1,3,5,... for the buccal group & 2,4,6,... for the vaginal group) to receive 400 microgram misoprostol.
  Interventions: Drug: Misoprostol (given buccally); Drug: Misoprostol (given vaginally)

INTERVENTIONS:
Drug: Misoprostol (given buccally) — 400 microgram misoprostol given buccally three hours before dilation and curettage (PHARMACIA CORPORATION - Istanbul, serial number 022-00, a tablet contains 200 micrograms)
  Other Names: serial number 022-00
  Arms: Buccal Misoprostol; Buccal and Vaginal Misoprostol
Drug: Misoprostol (given vaginally) — 400 microgram misoprostol (MISOPROSTOL - PHARMACIA CORPORATION - Istanbul, serial number 022-00, a tablet contains 200 micrograms)
  Other Names: serial number 022-00
  Arms: Buccal and Vaginal Misoprostol; Vaginal Misoprostol

SUMMARY:
The purpose of this study is to determine the effectiveness of buccal misoprostol and comparing this with vaginal route of the same drug.

ELIGIBILITY:
Inclusion Criteria:

* first trimester missed abortion

Exclusion Criteria:

* history or evidence of disorders that represent contraindication to the use of misoprostol:

  * severe pulmonary diseases
  * congenital or acquired heart diseases
  * glaucoma
  * prolonged use of corticosteroid
  * sickle cell anemia and adrenal insufficiency
  * smokers
  * known hypersensitivity to drugs
  * any evidence of infection
* patient's refusal to participate in the study
* patients with abnormal results of investigations
* patients with previous operations on cervix like conisation, cauterization, previous dilatation and curettage
* patients with complete abortion
* patients with severe bleeding that required emergency surgical evacuation of the uterus
* patients with partially dissolved tablets at the site of application in both groups

Ages: 19 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2007-03; Primary Completion 2008-01 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
To compare the efficacy of buccal administration to the more commonly vaginal route for preoperative cervical and priming in patients with first trimester surgical abortion. (Buccal Vs. Vaginal Misoprostol in the First Trimester Missed Abortion.) | March 2007 to March 2008

SECONDARY OUTCOMES:
The secondary objectives are to compare the side effects and acceptability by the subjects. | March 2007 to March 2008

CONTACTS AND LOCATIONS:
Overall Officials: BASHAR Y F HANOOSHI, CABOG, Principal Investigator — IRAQI MEDICAL SPECIALIZATION/IRAQ
Locations (1):
- Iraqi Medical Specialization, Risafa, Baghdad Governorate, Iraq